CLINICAL TRIAL: NCT02672670
Title: Effects of a Coping-oriented Supportive Programme (COSP) for People With Spinal Cord Injury During Inpatient Rehabilitation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, LI Yan, PhD student, The Hong Kong Polytechnic University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSEARS20151219002
Record Dates: First submitted 2016-01-20; First posted 2016-02-03 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Spinal Cord Injury; Psychosocial Problem
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Coping-oriented supportive programme (Experimental): Coping-oriented supportive programme: education of the SCI disease information, learning from role model by watching a well-established DVD, discussion about how to break down stressors and used appropriate coping strategies (problem-solving training, cognitive re-constructing, relaxation exercises, and activity scheduling) to manage the stressors relating to SCI. Social skills training and ways of maintaining and improving social support will also be discussed and practiced in the COSP.
  Interventions: Behavioral: Experimental: Intervention group---coping-oriented supportive programme
- A didactic group (Active Comparator): Usual rehabilitation care--routine inpatient rehabilitation care and brief education in groups (structured by both the rehabilitation nurses and the researcher), which will consist of similar professional contacts as the intervention (COSP) group, and thus can balance between the two study groups for the effect of social contacts and attention to SCI patients during group sessions. The intervention in the comparison group will be conducted by a rehabilitation nurse in the SCI wards. The knowledge/didactic education presented to the patients in the comparison group will be the basic health education and relevant information provided by the rehabilitation nurses in their routine care (mainly including knowledge of SCI, nutritional needs, skin care, bowel and bladder training, and other physical and psychological care of patients with SCI provided by the inpatient rehabilitation wards).
  Interventions: Behavioral: Active Comparator: Comparison group---a didactic talk (usual care)

INTERVENTIONS:
Behavioral: Experimental: Intervention group---coping-oriented supportive programme
  Other Names: COSP
  Arms: Coping-oriented supportive programme
Behavioral: Active Comparator: Comparison group---a didactic talk (usual care)
  Other Names: UC
  Arms: A didactic group

SUMMARY:
The aim of this proposed PhD study is to test the effectiveness of a newly developed coping-oriented supportive programme (COSP) for Chinese people with SCI during their early period of inpatient rehabilitation in Xi'an, China. The objectives of this study are to develop and validate the COSP in the inpatient rehabilitation hospitals; and to evaluate the effectiveness of this COSP for the SCI inpatients in two rehabilitation wards on their coping abilities, self-efficacy, mood status, and life satisfaction, when compared to those receiving routine care in another two rehabilitation wards. This proposed PhD study is a quasi-experimental study, using repeated-measures, comparison group design. The study will be conducted in two rehabilitation hospitals in Xi'an, China. There will be 50 patients in each of the two study groups (i.e., one intervention and one comparison group). The intervention group will receive the COSP including 8 weekly sessions, and the comparison group will receive usual rehabilitation care in brief didactic group-based education. Outcome measures will be examined at baseline and immediately, 1- and 3-month after completion of the interventions. The primary outcomes of this proposed study are coping ability and self-efficacy, while the secondary outcomes include mood status, life satisfaction, and pain. All data will be analysed using SPSS for Windows, version 21.0. Descriptive statistics will be employed for demographic and disease-related data and outcome scores. Data analysis for intervention effects will be based on both Per-protocol (PP) analyses and Intention-To-Treat (ITT). The missing data will be handled by the Last Observation Carried Forward (LOCF) strategy. Inferential statistics will be conducted for between-group and within-group comparison with specific considerations with the measurement level of the data and the fulfillment of the statistical assumptions of parametric or non-parametric tests, and further consider to use multivariate analysis of covariance (MANCOVA) or the analysis of covariance (ANCOVA).This study will provide evidence on the clinical effectiveness of the coping-oriented supportive programme in improving patients' psychological adjustment to SCI during earlier stage of inpatient rehabilitation, enhancing their psychosocial adaptation to the illness and subsequent life satisfaction and hence, integrating this psychosocial intervention into the conventional treatment and SCI rehabilitation practices.

ELIGIBILITY:
Inclusion Criteria:

* Planned to stay at the hospital for inpatient rehabilitation at least for three months;
* Traumatic injury or nontraumatic injury diagnosed by the physician, and within 2 years onset of the illness;
* Aged 18 to 64 years adults, able to communicate in Mandarin;
* Able to understand and follow the instructions and practices as required by the COSP programme;
* Voluntarily participating and with capacity to provide written or verbal consent.

Exclusion Criteria:

* Cognitively impaired (Mini Mental State Examination test score less than 23);
* Current mental illness (diagnosed as schizophrenia, anxiety disorder, or mood disorders), which can interfere with the understanding and learning provided by the intervention;
* Suffering from severe pain (NRS more than 7), frequent or much somatic complaints, social withdrawal as shown in the patient progressive sheets or physician's recent assessment records;
* High risk of self-harm (i.e., having a plan to hurt him/herself and having suicidal intention or ideas expressed recently);
* Currently engaged in another psychotherapeutic intervention(s) (e.g., psycho-education, social skills training, CBT, structured counseling programme, or other psychotherapies), and currently involved in any interventional trial.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-08; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Changes in coping ability (assessed by the Coping Orientations to Problems Experienced Inventory)during 3-month follow-up | Baseline, immediately after, 1- and 3-month post intervention
  This proposed study will need to have repeated measures to see the short-to-long term effects of the COSP by measuring the changes of participants' coping ability.
Changes in self-efficacy (assessed by the Moorong Self Efficacy Scale)during 3-month follow-up | Baseline, immediately after, 1- and 3-month post intervention
  This proposed study will need to have repeated measures to see the short-to-long term effects of the COSP by measuring the changes of participants' self-efficacy.

SECONDARY OUTCOMES:
Changes in mood (assessed by Hospital Anxiety and Depression Scale) during 3-month follow-up | Baseline, immediately after, 1- and 3-month post intervention
  This proposed study will need to have repeated measures to see the short-to-long term effects of the COSP by measuring the changes of participants' mood.
Changes in life satisfaction (assessed by Quality of Life Enjoyment and Satisfaction Questionnaire-Short Form) during 3-month follow-up | Baseline, immediately after, 1- and 3-month post intervention
  This proposed study will need to have repeated measures to see the short-to-long term effects of the COSP by measuring the changes of participants' life satisfaction.
Changes in Pain (assessed by the Numerical Rating Scale) during 3-month follow-up | Baseline, immediately after, 1- and 3-month post intervention
  This proposed study will need to have repeated measures to see the short-to-long term effects of the COSP by measuring the changes of participants' pain level.

CONTACTS AND LOCATIONS:
Locations (1):
- Yan LI, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No